CLINICAL TRIAL: NCT01175967
Title: Use of Palliative Performance and Symptom Distress Scales in Older Patients With Advanced Ovarian Cancer
Status: Terminated | Type: Observational
Why Stopped: Unable to meet accrual due to changing practice patters
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC1015; P30CA016086 (NIH); UNC-LCCC-1015
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Ovarian Cancer
Keywords: psychosocial effects of cancer and its treatment; perioperative/postoperative complications; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Postoperative Complications; Carcinoma, Ovarian Epithelial | interventions — Geriatric Assessment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Palliative Performance Scale version 2 (PPSv2) — PPSv2 is arrayed on a scaled from 10 (bedbound) to 100 (full ambulation) at 10 points increment. It will be administered beginning at baseline, post surgery (at the first post-operative clinic visit), 14-21 days post chemotherapy (post cycle 3 and post cycle 6), and at the first follow-up visit
Other: McCorkle Symptom Distress Scale (SDS) — A 13-item scale of SDS is used to indicate the degree of distress for a given symptom on a 5 point Likert Scale, ranging from 1 (least amount of distress) to 5 (extreme distress). This will be administered at baseline, post surgery (at the first post-operative clinic visit), 14-21 days post chemotherapy (post cycle 3 and post cycle 6), and at the first follow-up visit
Other: Geriatric Assessment — This will evaluate the subject's overall geriatric status. The first part will be filled out by the study team and the second half of the assessment will be populated with information provided by the subject. This will be completed at baseline, 2 weeks post-surgery and 14-21 days after completing cycle 3 and cycle 6.
Other: Medical Records Abstraction — Data collected from medical records will include information on surgical complications and chemotherapy toxicities, dose reductions, and any change in choice of chemotherapy drug. This will occur continuously throughout the study.

SUMMARY:
RATIONALE: Measuring changes in performance status and symptoms distress in patients with cancer may help doctors predict how patients will respond to treatment, and may help the study of cancer in the future.

PURPOSE: This clinical trial is studying changes in performance status and symptoms distress in older patients with advanced ovarian epithelial cancer undergoing surgery and/or chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the changes in performance status and symptom distress in older patients with presumed or advanced ovarian cancer undergoing surgery and/or chemotherapy.

Secondary

* To explore the association between these changes with chemotherapy drug change, dose reduction, or dose delay due to toxicity in these patients.
* To explore the association between these changes with the development of surgical complications in these patients.
* To observe the response in the Geriatric Assessment (GA) and report the individual item scores.

OUTLINE: Patients complete the Palliative Performance Scale and the McCorkle Symptom Distress Scale questionnaires at baseline, at 10-20 days after surgery*, at 14-21 days after courses 3 and 6 of chemotherapy ( if applicable), and at approximately 2-3 months at the patient's first follow-up visit. The research team completes the Professional Geriatric Assessments. Patients' medical records are also reviewed for any surgical complications, chemotherapy toxicities, dose reductions or delays, or change in medications secondary to chemotherapy toxicities.

NOTE: *Patients who complete the assessments and questionnaires at baseline but who are found not to have ovarian cancer during surgery will remain eligible for assessment of surgical complications.

ELIGIBILITY:
Inclusion Criteria:

* Clinical findings highly suggestive of advanced ovarian epithelial cancer undergoing surgery for definitive diagnosis and staging
* ≥ 65 years of age

Exclusion Criteria:

* Prior diagnosis of ovarian cancer
* Inability to read and speak English
* Inability to comply with study requirements

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who undergo surgery for presumed ovarian cancer, and those diagnosed with ovarian cancer who undergo surgery and chemotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Changes in scale score after surgery and/or chemotherapy | baseline, post surgery (at the first post-operative clinic visit), 14-21 days post chemotherapy (post cycle 3 and post cycle 6), and at the first follow-up visit
  Results will be described by scoring outcome from a professional assessment of performance status as measured by PPSv2, and from a SDS survey which asks about the perceived level of symptom distress the patient is experiencing.PPSv2 is arrayed on a scaled from 10 (bedbound) to 100 (full ambulation) at 10 points increment. A 13-item scale of SDS is used to indicate the degree of distress for a given symptom on a 5 point Likert Scale, ranging from 1 (least amount of distress) to 5 (extreme distress)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Van Le, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States